CLINICAL TRIAL: NCT05083728
Title: An Observational Study of Calibrated CT Scans to Evaluate Shoulder Geometry and Bone Density for Finite Element Analysis (FEA) on a Simulated Surgical Implant
Brief Title: S-32 PG 242 Short Stem
Status: Completed | Type: Observational
Sponsor: St. Louis Joint Replacement Institute (Other)
Collaborators: Lima Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21-06-2182
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2021-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT — Clinicians are free to choose the adult subjects in whom a non-contrast calibrated CT-scan will be performed as a part of routine clinical care. The decision to order a noncontrast CT-scan of the shoulder must be made prior to, and independently from, the decision to enroll the patient.

SUMMARY:
The data of calibrated CT-scans will be used for the Finite Element Analysis (FEA) analysis for SMR Short Stem in identified hospitals in EU and US as developers of the project and for further research, upon subject acceptance.

In particular, the Quantitative Computer Tomography (QTC)/Finite Element Analysis (FEA) model of the assembly consisting of the shoulder and the orthopaedic implant allows detailed analyses including:

* assessment of micromotion at the bone-implant interface, to predict osseointegration;
* comparison of strains/stresses between the intact bone tissue and the bone with the implant in order to predict the stress shielding phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects (males and/or females) must be ≥ 18 years of age

  2. Subjects are willing and able to provide written informed consent for collection of the data; if a patient has already completed and performed the calibrated CT-scans as per standard clinical practice, the subject may be contacted to offer participation in the study.

  3. Adult patients who will undergo noncontrast CT scanning of the shoulder as part of routine preoperative planning for shoulder arthroplasty will be eligible to participate in the study and receive a calibrated CT scan of the shoulder. The decision to undergo CT scan will be made independently of study participation; only patients who require a CT scan of the shoulder for clinically necessary reasons are eligible to participate.

Exclusion Criteria:

* 1. Pregnancy or lactation; 2. Subjects who have fracture of the affected shoulder; 3. Subjects who have had prior surgery on the affected shoulder that resulted in metal implants, including but not limited to:
* Partial or total shoulder joint replacement;
* Open reduction internal fixation of fracture;
* Prior rotator cuff repair with metal implants; 4. Local or systemic infection; 5. Persistent acute or chronic osteomyelitis; 6. Focal vascular or neurologic diseases affecting the concerned limb; 7. Metabolic disorders or systemic diseases that substantially affect bone quality, including the following:
* Renal osteodystrophy
* Osteoporosis
* Osteomalacia
* Osteopetrosis 8. Bone tumors involving the shoulder girdle; 9. Local or disseminated neoplastic diseases; 10. Severe deformity including malunion, nonunion, excessive bone loss that would result in improper virtual implant positioning;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible patient population for this study will include all patients who require a noncontrast CT as a part of their clinical care. The effective number of cases included will depend on the availability and quality of calibrated CT-scan imaging data necessary to perform FEA as detailed in the selection criteria.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Collection of calibrated CT scans to obtain human imaging data to perform a Finite Element Analysis (FEA) on a simulated surgery using a specific implant, as per clinical practice. | <24 hours
  To perform the Finite Element Analysis (FEA), the following data will be requested:
  * Shoulder calibrated CT-scan
  * Date of calibrated CT-scan execution
  * Subject's year of birth
  * Subject's sex
  * Subject's weight
  * Subject's height
  * Subject's ethnicity

CONTACTS AND LOCATIONS:
Locations (1):
- SSM Health- DePaul, Bridgeton, Missouri, United States